CLINICAL TRIAL: NCT00064883
Title: The Natural History of Childhood Malignancies Treated With Radiation Therapy
Brief Title: Radiation Therapy and the Natural History of Childhood Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030241; 03-C-0241; NCT00068536 (obsolete NCT alias)
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Cancer; Childhood Malignancy
Keywords: Radiation Therapy; Children; Cancer; Late Effects; Natural History; Radiation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Pediatric cancer patients referred to the ROB who have received or require radiation therapy

SUMMARY:
This study will: 1) provide standard non-experimental radiation therapy to children who have a form of cancer or similar disease process that is of scientific interest, importance, or educational value; 2) determine the effects of radiation on childhood cancers; and 3) allow for the education of nurses, medical students, residents, clinical fellows, and physicians in the management and care of this specialized group of cancer patients. Patients in this study will not receive experimental therapy, but will be given standard medical care.

Patients eligible for this study include: 1) children with cancer or a precancer syndrome, such as aplastic anemia or other myelodysplastic syndrome, who are between 3 years and 21 years of age and whose disease will be treated or has been treated with radiation therapy in the NCI's Radiation Oncology Branch (ROB); 2) patients with cancer or a precancer syndrome who have disease manifestations of special interest to ROB investigators; and 3) patients with cancer or a precancer syndrome who offer an important educational benefit to radiation oncology trainees and staff.

Participants will undergo a medical history, physical examination, and blood tests, and radiation therapy. Before beginning treatment, medical information such as pathology reports, laboratory results, diagnosis and treatment history, scan results, and so forth, will be obtained from the patient's medical records. Additional procedures that may need to be done include scans, such as magnetic resonance imaging (MRI), computed tomography (CT), positron emission tomography (PET), lung function tests, arteriogram, or tumor biopsies.

Participants will then have a (simulation) treatment planning session for radiation therapy during which measurements are taken, CT images are taken, and markings are placed on the body to help determine the treatment area. The radiation will be delivered to the body by a machine called a linear accelerator, which produces x-rays. Radiation therapy is generally given once or twice a day 5 days a week. Each treatment takes about 10 minutes.

When the course of treatment is completed, patients return to the Radiation Oncology clinic for follow-up visits that include blood tests, a physical examination, and review of symptoms, if any. Visits are kept to a minimum, but continue for a prolonged period to watch for any late effects of treatment that may occur over a period of decades.

DETAILED DESCRIPTION:
BACKGROUND

-Children with cancer represent relatively rare disorders that are of unique scientific importance and educational value.

OBJECTIVE

-This protocol will allow follow-up of these patients for determination of the effects of radiation on overall survival, as well as relapse-free/ disease-free survival, local control, and the late sequelae of radiation therapy.

ELIGIBILITY

-Children with cancer and who require radiation are referred to the Radiation Oncology Branch primarily from Children's National Medical Center in Washington, D.C. and from other Branches of the NCI/NIH.

DESIGN

-This protocol is designed to provide the radiation component of therapy in children with cancer that have diseases that are of unique scientific interests, importance, and/or educational value.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who are evaluated by the Radiation Oncology Branch and are:

Children with cancer (or a precancer syndromes, such as aplastic anemia or other myelodysplastic syndromes), between the age(s) of 3 - 21 years, whose cancer (or precancer syndrome) will be treated with radiation therapy in the Radiation Oncology Branch, NCI.

Patients with cancer (or a precancer syndromes, such as aplastic anemia or other myelodysplastic syndromes), who present with disease manifestations of special interest to Radiation Oncology Branch investigators, because they are likely to shed led light on the natural history, pathogenesis, radiation response, and late effects of disease process.

Patients with cancer (or precancer syndromes, such as aplastic anemia or other myelodysplastic syndromes) who offer an important educational benefit to trainees in radiation oncology and staff.

Patient must have a primary physician in the community who specializes in pediatrics and/or oncology and is willing to collaborate with the ROB staff in the clinical management of the patient

If indicated, availability of a parent or legal guardian to give informed consent

Children with cancer (or a precancer syndrome, such as aplastic anemia or other myelodysplastic syndrome), between the age(s) of 3- 21 years, whose cancer (or precancer syndrome) have already been treated with radiation therapy in the Radiation Oncology Branch, NCI.

EXCLUSION CRITERIA:

Patients, and/or guardians who are in the estimation of the PI, deemed unable or unlikely to adhere to protocol treatment and follow-up requirements.

Patients who are enrolled on a clinical trial (e.g. COG or CNMC) in which one of the research objectives is to study the radiation treatment.

Patients who are pregnant and are to receive radiation treatment on this protocol.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cancer (or a precancer syndrome, such as aplastic anemia or other myelodysplastic syndrome) who require radiation
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2003-07-28 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in patient disease after radiation | at completion of treatment
  Overall response

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-C-0241.html